CLINICAL TRIAL: NCT05078658
Title: Low-carbohydrate Diet in Paediatric Type 1 Diabetes: Effects on Glycaemic Control and Islet Autoimmunity
Brief Title: Low-carbohydrate Diet in Children with Type 1 Diabetes
Acronym: Lowca
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Collaborators: Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Zdeněk Šumník, Prof., University Hospital, Motol
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NU21-01-00085
Record Dates: First submitted 2021-09-15; First posted 2021-10-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-carbohydrate diet (Experimental): The subjects will be delivered five pre-made ready meals per day throughout the period (5 weeks). These will contain age- and gender-specific recommended amount of calories but the amount of carbohydrates would be limited to provide only 15% (+/- 5%) of the recommended energy a day.
  Interventions: Other: Low-carbohydrate diet
- Recommended carbohydrate diet (Active Comparator): The subjects will be delivered five pre-made ready meals per day throughout the period (5 weeks). These will contain age- and gender-specific recommended amount of calories with 50% (+/- 5%) of the recommended energy from carbohydrates.
  Interventions: Other: Recommended-carbohydrate diet

INTERVENTIONS:
Other: Low-carbohydrate diet — The diet will contain age- and gender-specific recommended amount of calories but the amount of carbohydrates would be limited to provide only 15% (+/- 5%) of the recommended energy a day.
  Arms: Low-carbohydrate diet
Other: Recommended-carbohydrate diet — The subjects will be delivered five pre-made ready meals per day throughout the period (5 weeks). These will contain age- and gender-specific recommended amount of calories with the amount of carbohydrates equal to 45% (+/- 5%) of the recommended energy a day.
  Arms: Recommended carbohydrate diet

SUMMARY:
The primary aim of this pilot study is to test whether low-carbohydrate diet (LCD) instituted in children/adolescents with type 1 diabetes (T1D) can improve their disease control. The primary objective of the trial is the change in continuous glucose monitoring time in target range 3.9-10.0 mmol/l (TIR) in a 5-week period on LCD as opposed to a 5-week period on recommended carbohydrate diet (RCD).

Secondary objectives are:

Changes in immune parameters during the LCD period; Differences in fecal microbiome during the LCD period; Differences in fecal, serum and urine metabolome during the LCD period;

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosed according to the ADA (American Diabetes Assocciation) criteria
* T1D duration for at least 1 year prior to the intervention
* continuous glucose monitor (CGM) worn > 70% time in the month prior to the intervention

Exclusion Criteria:

* last HbA1c < 40 or > 70 mmol/mol
* subject has celiac disease
* daily average carbohydrate intake < 130 g/day from 14 days food record prior to the intervention
* any concomitant disease possibly affecting glucose control
* any chronic medication possibly affecting glucose control

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in continuous glucose monitoring time in target range (3.9-10.0 mmol/l) during the LCD period compared to the RCD period | Month 1 - Month 24

SECONDARY OUTCOMES:
Changes in mean insulin dose during the LCD period compared to the RCD period | Month 1 - Month 24
Changes in mean body weight standard deviation score during the LCD period compared to the RCD period | Month 1 - Month 24
Changes in the lipid spectrum during the LCD period compared to the RCD period | Month 1 - Month 24
Changes in muscle strength measured by jumping mechanography during the LCD period compared to the RCD period | Month 1 - Month 24
Changes in lymphocyte subgroup cell counts (flow cytometry) during the LCD period | Month 1 - Month 36
Differences in faecal microbiome between the LCD and RCD periods | Month 1 - Month 36
Differences in faecal metabolome between the LCD and RCD periods | Month 1 - Month 36
Differences in serum metabolome between the LCD and RCD periods | Month 1 - Month 36
Differences in urine metabolome between the LCD and RCD periods | Month 1 - Month 36

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Motol, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No